CLINICAL TRIAL: NCT02755103
Title: Mindfulness Meditation for the Treatment of Women With Comorbid PTSD and SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Therese K. Killeen, Research Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00048115; R01DA040968 (NIH)
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Results first posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Stress Disorders, Post-Traumatic; Substance-Related Disorders
Keywords: Mindfulness; Comorbid PTSD and SUD; Meditation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Women receiving MBRP plus TAU (Experimental): Women will receive the Mindfulness Based Relapse Prevention (MBRP) plus treatment as usual (TAU less trauma focused group).
  Interventions: Behavioral: Mindfulness Based Relapse Prevention (MBRP)
- Women receiving TAU (No Intervention): Women will only receive treatment as usual (TAU less trauma focused group).

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention (MBRP) — MBRP integrates coping skills from cognitive-behavioral relapse prevention therapy with Mindfulness Meditation (MM) practices, raising awareness of substance use triggers and reactive behavioral patterns, and teaching skillful coping responses.
  Arms: Women receiving MBRP plus TAU

SUMMARY:
The current study will modify an already existing therapy for individuals with substance use disorders to address Post Traumatic Stress Disorder (PTSD) in women enrolled in substance use disorders (SUD) treatment who suffer with both PTSD and SUD. Mindfulness meditation has been shown to help individuals to cope with stress and regulate emotions. Through meditation practice women will experience less distress related to PTSD symptoms and reduced substance use in response to emotional triggers. Women enrolled in intensive SUD treatment at a community program will be randomized to receive either 8 weeks of 90 minute Mindfulness Based Relapse Prevention (MBRP) group sessions plus treatment as usual (TAU) or TAU alone. The MBRP group sessions will replace 90 minutes of TAU group therapy. Measures of feasibility of implementation, acceptance and adherence will be obtained. Preliminary efficacy for substance use and PTSD symptom severity will be measured at post treatment and at 3- and 6- months' follow-up.

DETAILED DESCRIPTION:
This randomized controlled pilot study will evaluate the feasibility and preliminary efficacy of MBRP plus usual community treatment as usual (TAU) compared to TAU alone (TAU) for women with substance use disorders(SUD) and PTSD enrolled in community substance abuse treatment. Participants will be randomized to eight weekly 90-minute, mixed individual and group-based MBRP in addition to TAU or TAU alone. The eight sessions of MBRP will replace 8 sessions of seeking safety (SS); a trauma focused integrated therapy currently implemented in TAU. Outcomes assessed will be:

1. PTSD symptom severity as measured by the Clinician's Administered PTSD Scale (CAPS) and Post Traumatic Stress Disorder Symptom Scale-Self Report (PSS-SR);
2. Alcohol and substance use as measured by the Timeline Follow Back (TLFB) assessment and corroborated with urine drug screens.
3. psychosocial functioning;
4. Measure of emotional regulation and mindfulness awareness, attention and acceptance.

Recruitment of participants will primarily take place a community treatment program treating women with co-occurring PTSD and SUD.

Following therapist training, certification and piloting, eligible women will be invited to participate in the study. Interested potential participants will be screened for major inclusion/exclusion criteria including age, alcohol/substance use, history of trauma and psychiatric/health/medication status. If potentially eligible, an Institutional Review Board (IRB) approved informed consent will be obtained and participants will be scheduled for a baseline assessment appointment. If an individual is ineligible to participate in this research protocol, she will continue in her usual community treatment program and/or if indicated, be referred for additional treatment services. The investigators decided to limit the study group to women because they represent the largest percentage of patients with comorbid PTSD and SUDs and most have experienced sexual and/or physical trauma. So when trauma-focused treatment is delivered in a group setting for this population, single sex groups create a safe, comfortable and open atmosphere that is required for MM-based treatment and trauma focused work. After having at least 7 days in standard treatment baseline assessments will be collected. Women meeting inclusion with no exclusionary criteria will be randomized to MBRP plus TAU or TAU alone control. Both groups will attend their standard intensive TAU program. The eight MBRP therapy sessions will be integrated into the standard TAU program and replace 8 TAU SS sessions. Participants will be introduced to the therapists and scheduled for their first individual/small group session.

The primary outcome measures for the efficacy portion of this study are 1) the effective reduction in PTSD symptom severity through the total score on the CAPS at the end of treatment between the two study groups and 2) the effective reduction in the proportion of days using and amount of use of alcohol/substances during the final 30 days of treatment as measured by the TLFB verified by urine drug screens (UDS). In addition, secondary endpoints will include CAPS scores at the 3 and 6 month post-intervention follow-up visits, the 7 day point prevalence abstinence rates at each treatment, post treatment and follow up visits. Also, PSS-SR, Obsessive Compulsive Drinking and Substance Use Scale-Revised (OCDS-R), Addiction Severity Index-Lite (ASI-Lite), Difficulties in Emotional Regulation Scale (DERS), Mindfulness Acceptance and Awareness Questionnaire (MAAS), Five Facet Mindfulness Questionnaire (FFQS) and Cognitive and Affective Regulation Scale (CAMS-R). There will also be secondary endpoints and used to gain insight into potential effect modification and mediation. Secondary analysis will also include the proportion of days using alcohol/drugs, craving, psychosocial functioning and emotional regulation. Participants will be assessed weekly throughout the intervention, at the end of the intervention and at 3- and 6- month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 65 years of age enrolled in the Charleston Center (CC) intensive outpatient and New Life program treatment.
* Able to comprehend English.
* Meets fifth edition Diagnostic and Statistical Manual V (DSM V) criteria for current alcohol or substance use disorder and have used alcohol/substances in the 30 days prior to clinic treatment entry.
* Meets DSM V criteria for current PTSD with a score greater than or equal to 25 on the CAPS 5.0.
* Participants may also meet criteria for a mood or anxiety disorder. Participants on psychotropic medications for a mood or anxiety disorder must have been stabilized on medications for at least 4 weeks before therapy initiation.
* Able to adequately provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
* Willing to commit to 8 therapy sessions, baseline, weekly and follow-up assessments.

Exclusion Criteria:

* Current primary psychotic or thought disorder (i.e. Schizophrenia or schizoaffective disorder, mania), major depression with suicidal ideation, dissociative identity disorder and/or homicidal ideations.
* Present a serious suicide risk, such as those with severe depression, or who are likely to require hospitalization during the course of the study.
* In ongoing therapy for PTSD either within or outside of the CC, who are not willing to discontinue these therapies for the duration of the study therapy,
* Unstable medical condition or one that may require hospitalization during the course of the study.
* Women who are pregnant or planning to become pregnant.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Therese K Killeen, PhD APRN, Principal Investigator — Medical University of South Carolina
Locations (1):
- The Charleston Center, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Killeen TK, Wen CC, Neelon B, Baker N. Predictors of Treatment Completion among Women Receiving Integrated Treatment for Comorbid Posttraumatic Stress and Substance Use Disorders. Subst Use Misuse. 2023;58(4):500-511. doi: 10.1080/10826084.2023.2170183. Epub 2023 Jan 27. PMID 36705433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Started | 45 | 45
8 Week Follow-up Completed | 32 | 28
3 Month Follow-up Completed | 26 | 27
Completed (6 Month Follow-up Completed) | 25 | 27
Not Completed | 20 | 18
Not completed — Lost to Follow-up | 17 | 15
Not completed — Death | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (9.2) | 32.1 (6.1) | 32.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 45 | 90
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 42 | 42 | 84
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 13 | 21
  White | 31 | 26 | 57
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90
Clinician Administered Posttraumatic Stress Disorder Scale - 5 (CAPS-5) [Mean (Standard Deviation); unit: Scores on a scale] — The Clinician-Administered Post Traumatic Stress Disorder Scale (CAPS-5) is a 20 item structured interview that assesses the frequency and severity of Post Traumatic Stress Disorder (PTSD) symptoms on a scale of 0 (absent) to 4 (extreme/incapacitating). Participants are asked to rate the frequency and severity of the symptoms they are experiencing. Scores are summed for a total score and higher scores represent higher symptom severity. Score range is 0-80. Mean baseline total scores are reported here.
  Scores on a scale | 42 (10) | 41 (10.4) | 41.5 (10.1)
Post Traumatic Stress Symptom Severity Scale- Self Report [Mean (Standard Deviation); unit: Scores on a scale] — Post Traumatic Symptom Severity Self Report (PSS-SR) is a 17-item self-reported questionnaire to assess symptoms of Post Traumatic Stress Disorder. Three questions representing new Diagnostic and Statistical Manual 5 (DSM5) criteria for Post Traumatic Stress Disorder were added. The 20 items describe symptom frequency and severity on a scale ranging from 0 (not at all or only one time) to 3 (almost always or five or more times per week). Higher scores represent greater symptom severity and worsening of symptoms. The range of scores is 0 - 60. Mean baseline total scores are reported here.
  Scores on a scale | 34.1 (12.8) | 32.8 (12.9) | 33.4 (11.3)
Time Line Follow Back [Count of Participants; unit: Participants] — The Time Line Follow Back (TLFB) is an interview using a calendar method to prompt recall of any use of alcohol and/or other substances including cannabis, stimulants, opioids, cocaine and sedatives over a given period of time. Participants are asked to recall the number of days they used alcohol and/or other substances such that the percent days using over a given period of time can be calculated. The baseline time period represents 60 days prior to enrollment.
  Participants
    Any alcohol use | 25 | 28 | 53
    Any cannabis use | 14 | 25 | 39
    Any stimulant use | 15 | 13 | 28
    Any opioid use | 19 | 18 | 37
    Any cocaine use | 15 | 15 | 30
    Any sedative use | 4 | 6 | 10
Time Line Follow Back [Mean (Standard Deviation); unit: percentage of days] — The Time Line Follow Back (TLFB) is an interview using a calendar method to prompt recall of frequency of alcohol and/or other substance use including cannabis, stimulants, opioids, cocaine and sedatives over a given period of time. Participants are asked to recall the number of days they used alcohol and/or other substances such that the percent days using over a given period of time can be calculated.The time period for the baseline interview is 60 days prior to enrollment.
  percentage of days
    Percent alcohol drinking days | 40.9 (38.9) | 48.5 (40.3) | 44.9 (39.4)
    Percent cannabis use days | 58.9 (41.6) | 55.7 (41.6) | 56.8 (41.1)
    Percent stimulant use days | 41.6 (38.3) | 54.4 (41.4) | 47.5 (39.5)
    Percent opioid use days | 77.5 (36.5) | 80.6 (31.3) | 79.1 (33.6)
    Percent cocaine use days | 57.1 (37) | 50.8 (42.4) | 53.9 (39.2)
    Percent sedative use days | 49.2 (36.5) | 56.8 (45.7) | 54.8 (40.3)
Difficulty in Emotional Regulation (DERS) [Mean (Standard Deviation); unit: Scores on a scale] — The Difficulty in Emotion Regulation Scale (DERS) is a 36-item self-report measure developed to assess clinically significant difficulties in emotion regulation. Responses range from 1 (almost never) to 5 (almost always) with higher scores indicating greater difficulties in emotion regulation. The range of scores is 0 to 180 and item scores are summed for a total score. Mean baseline total scores are reported here.
  Scores on a scale | 105.6 (28.8) | 101.1 (28.8) | 103.3 (29.4)
Five Factor Mindfulnes Questionaire (FFMQ) [Mean (Standard Deviation); unit: Scores on a scale] — The Five Factor Mindfulness Questionnaire (FFMQ) is a 24 item self report scale that measures the trait-like tendency to be mindful in daily life. It is comprised of aspects of mindfulness such as observing, describing, acting with awareness, non-judging, and non-reactivity. Item ratings range from 1 (never or very rarely true) to 5 (very often true or always true) and items are summed for a total score. Higher scores represent higher levels of mindfulness. Mean baseline total scores are reported here.
  Scores on a scale | 71.6 (16.1) | 72.7 (16.1) | 72.1 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered Posttraumatic Stress Disorder Scale for DSM-5
Description: The Clinician-Administered Post Traumatic Stress Disorder Scale fifth edition (CAPS-5) is a 20 item structured interview that assesses the frequency and severity of Post Traumatic Stress Disorder (PTSD) symptoms on a scale of 0 (absent) to 4 (extreme/incapacitating). Scores are summed for a total score and higher scores represent higher symptom severity. Score range is 0-80.
Time Frame: 8 weeks (60 days baseline to end of treatment). Missing scores were imputed. Scores presented are controlled for baseline scores.
Population: Mean scale scores for participants at the end of treatment (baseline to end of treatment).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 45 | 45
score on a scale | 16.5 (2.3) | 18.5 (2.4)

2. Secondary Outcome: Clinician Administered Posttraumatic Stress Disorder Scale-5 (CAPS-5)
Description: The Clinician-Administered Post Traumatic Stress Disorder Scale fifth edition (CAPS-5) is a 20 item structured interview that assesses the frequency and severity of Post Traumatic Stress Disorder (PTSD) symptoms on a scale of 0 (absent) to 4 (extreme/incapacitating). Scores are summed for a total score and higher scores represent higher symptom severity. Score range is 0-80. Group differences in PTSD symptom severity are reported here.
Time Frame: 3 (90 days from end of treatment to 3 month follow-up) and 6 (90 days from 3 month follow-up to 6 month follow-up) month follow-up. Missing scores are imputed. Scores presented are controlled for baseline scores.
Population: Mean scores for participants at 3 and 6 month follow-up visits. Missing data scores were imputed. Scores presented are controlled for baseline scores.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 45 | 45
score on a scale
  3 month follow-up | 13.8 (2.4) | 16.1 (2.4)
  6 month follow-up | 12.7 (2.5) | 13.3 (2.5)

3. Secondary Outcome: Post Traumatic Stress Disorder Symptom Scale- Self Report (PSS-SR)
Description: Post Traumatic Symptom Severity Self Report (PSS-SR) is a 17-item self-reported questionnaire to assess symptoms of Post Traumatic Stress Disorder. Three questions representing the three new Diagnostic and Statistical Manual 5 (DSM5) criteria for Post Traumatic Stress Disorder were added. Each of the 20 items describe Post Traumatic Stress Disorder symptoms which participants rate in terms of their frequency or severity using a Likert-type scale ranging from 0 (not at all or only one time) to 3 (almost always or five or more times per week). Higher scores represent greater symptom severity and worsening of symptoms. The range of scores is 0 - 60.
Time Frame: weekly during treatment, end of treatment 8 weeks, 3 and 6 month follow-up. Missing scores were imputed at different time periods. Scores presented are controlled for baseline scores.
Population: Mean total Post Traumatic Symptom Severity Self Report (PSS-SR) scores for participants throughout the study period. Missing scores were imputed at different time periods. Scores presented are controlled for baseline scores.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 45 | 45
score on a scale
  Week 1 | 30.6 (1.8) | 29.2 (1.8)
  Week 2 | 24.7 (1.8) | 28.3 (1.9)
  Week 3 | 24 (1.9) | 28.5 (2)
  Week 4 | 21.2 (1.9) | 24.3 (2)
  Week 5 | 17.9 (2.0) | 20.2 (2.1)
  Week 6 | 16 (2) | 20.3 (2.1)
  Week 7 | 16.7 (2.1) | 20 (2.2)
  Week 8 | 17.4 (2) | 18.4 (2.1)
  3 month follow-up | 15.6 (2.1) | 17.2 (2.1)
  6 month follow-up | 11.5 (2.2) | 19 (2.1)

4. Secondary Outcome: Time Line Follow Back (TLFB)
Description: The Time Line Follow Back (TLFB) is a calendar based interview method to prompt recall of frequency of drinking alcohol and/or using substances over a given time period. Participants are asked to report any days in which they used alcohol and/or other substances (cannabis, stimulants,opioids, cocaine, sedatives) during a given time period. The mean percent of days reporting use of alcohol (Percent Days Drinking:PDD) and/or substances ( Percent Days Using Substances:PDU) for those individuals who attended the end of study visit (n=60) and reported any use during treatment is reported here. The time period includes the 8 weeks from baseline to end of the treatment intervention.
Time Frame: 8 weeks (60 days from baseline to end of treatment).
Population: The mean percent days reporting use of alcohol and/or other substances (cannabis, stimulants, opioids, cocaine and sedatives) for those individuals who attended the end of treatment study visit (n=60) and reported any use during treatment. Those individuals who did not use alcohol or substances during treatment are not reported here. Different number of participants reported use of various different substances during treatment.
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 32 | 28
percent of days
  PDD 8 weeks: number analyzed (Participants) | 13 | 13
  PDD 8 weeks | 11 (.11) | 10 (.1)
  PDU cannabis 8 weeks: number analyzed (Participants) | 5 | 9
  PDU cannabis 8 weeks | 8 (.08) | 15 (.27)
  PDU stimulants 8 weeks: number analyzed (Participants) | 1 | 1
  PDU stimulants 8 weeks | 11 (.0) | 2 (.0)
  PDU opioids 8 weeks: number analyzed (Participants) | 3 | 0
  PDU opioids 8 weeks | 23 (.21) |
  PDU cocaine 8 weeks: number analyzed (Participants) | 3 | 3
  PDU cocaine 8 weeks | 18 (.28) | 4 (.02)
  PDU sedatives 8 weeks: number analyzed (Participants) | 4 | 1
  PDU sedatives 8 weeks | 1.6 (.005) | 1.4 (0)

5. Secondary Outcome: Time Line Follow Back (TLFB)
Description: The Time Line Follow Back (TLFB) is an interview using a calendar based method to prompt recall for frequency of alcohol and substance (cannabis, stimulants, opioids, cocaine and sedatives) use over a given time period. Participants are asked to report any days in which they used alcohol and/or other substances (cannabis, stimulants,opioids, cocaine, sedatives) during a given time period. The mean percent of days reporting use of alcohol (PDD) and/or substances (PDU: cannabis, stimulants, opioids, cocaine and sedatives) for those who attended the 3 month follow-up visit (n=53) and reported use of any alcohol and substances at the 3 month follow-up visit is reported here.
Time Frame: 3 month follow-up mean percent days using alcohol (PDD) and/or substances (PDU: cannabis, stimulants, opioids, cocaine and sedatives) for those who attended (n=53) and reported any use at the 3 month follow-up (90 days from 3 to 6 month) visit.
Population: Mean of percent days reporting use of alcohol and/or substances (cannabis, stimulants, opioids, cocaine and sedative) for those participants who attended the 3 month follow-up visit (n=53) and reported any alcohol and/or substance use at the 3 month follow-up visit. Those participants who did not report any alcohol and/or substance use are not represented here. Different number of participants reported use of various different substances at the 3 month follow-up visit.
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 26 | 27
percent of days
  PDD alcohol 3 month follow-up: number analyzed (Participants) | 8 | 10
  PDD alcohol 3 month follow-up | 21 (.28) | 15 (.14)
  PDU cannabis 3 month follow-up: number analyzed (Participants) | 6 | 6
  PDU cannabis 3 month follow-up | 26 (.4) | 21 (.17)
  PDU stimulants 3 month follow-up: number analyzed (Participants) | 1 | 3
  PDU stimulants 3 month follow-up | 10 (0) | 38 (.41)
  PDU opioids 3 month follow-up: number analyzed (Participants) | 2 | 2
  PDU opioids 3 month follow-up | 48 (.11) | 39 (.21)
  PDU cocaine 3 month follow-up: number analyzed (Participants) | 3 | 4
  PDU cocaine 3 month follow-up | 43 (.4) | 9 (.12)
  PDU sedatives 3 month follow-up: number analyzed (Participants) | 0 | 1
  PDU sedatives 3 month follow-up |  | 24 (0)

6. Secondary Outcome: Time Line Follow Back (TLFB)
Description: The Time Line Follow Back (TLFB) is an interview using a calendar based method to prompt recall for obtaining frequency of alcohol and/or substance (cannabis, stimulants, opioids, cocaine and sedatives) use over a given time period. Participants are asked to report any days in which they used alcohol and/or other substances (cannabis, stimulants,opioids, cocaine, sedatives) during a given time period. The mean percent of days reporting use of alcohol (PDD) and/or substances (PDU: cannabis, stimulants, opioids, cocaine and sedatives) for those who attended the 6 month follow-up visit (n=52) and reported any use of alcohol and/or substances at the 6 month follow-up visit is reported here.
Time Frame: 6 month follow-up mean percent days using alcohol (PDD) and/or substances (PDU: cannabis, stimulants, opioids, cocaine and sedatives) for those who attended (n=52) and reported any use at the 6 month follow-up (90 days from 3 to 6 month follow-up) visit.
Population: Mean percent days of use for participants attending (n=52) the 6 month follow-up visit and who reported use of alcohol and/or substances (cannabis, stimulants, opioids, cocaine and sedatives) at the 6 month follow-up visit. Individuals who did not report use of any alcohol and/or substances are not reported/represented here. Different number of participants reported use of various different substances at the 6 month follow-up visit.
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 25 | 27
percent of days
  PDD alcohol 6 month follow-up: number analyzed (Participants) | 7 | 13
  PDD alcohol 6 month follow-up | 9 (.11) | 21 (.22)
  PDU cannabis 6 month follow-up: number analyzed (Participants) | 4 | 7
  PDU cannabis 6 month follow-up | 18 (.27) | 17 (.25)
  PDU stimulant 6 month follow-up: number analyzed (Participants) | 0 | 4
  PDU stimulant 6 month follow-up |  | 3 (.01)
  PDU opioids 6 month follow-up: number analyzed (Participants) | 0 | 0
  PDU cocaine 6 month follow-up: number analyzed (Participants) | 3 | 2
  PDU cocaine 6 month follow-up | 1 (.16) | 27 (.16)
  PDU sedatives 6 month follow-up: number analyzed (Participants) | 0 | 1
  PDU sedatives 6 month follow-up |  | 1

7. Secondary Outcome: Time Line Follow Back (TLFB)
Description: Time Line Follow Back (TLFB) is a calendar based method that allows a clinician to get a quantitative amount of an individual's daily drinking during a given period of time. Participants are asked about the number of drinks they consumed on the days that they drank. The mean number of standard alcohol drinks per drinking day (DDD) for those individuals who reported any drinking days during treatment from baseline to end of treatment (n=26) is reported.
Time Frame: 8 weeks (60 days from baseline to end of treatment). Only those participants who reported any drinking at the are included (n=26). Those who did not report any alcohol use are not represented/reported here.
Population: Number of drinks per drinking day for participants who attended the 8 week end of study visit and used alcohol during the 8 weeks of treatment (n=26). Those individuals who did not report alcohol use are not reported here.
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 13 | 13
drinks per drinking day | 2.9 (2.4) | 2.5 (2.3)

8. Secondary Outcome: Time Line Follow Back (TLFB)
Description: Time Line Follow Back (TLFB) is a calendar based method that allows a clinician to obtain a quantitative amount of an individual's daily drinking during a given period of time. Participants are asked about the number of drinks they consumed on the days that they drank.The mean number of standard alcohol drinks per drinking day (DDD) for those individuals who reported any drinking from the end of treatment to the 3 month follow-up visit (n=18) is reported.
Time Frame: 3 month follow-up (90 days from end of treatment to 3 month follow-up). Only those participants who reported any drinking at the 3 month follow-up visit (n=18) are included.
Population: 3 months follow-up mean drinks per drinking day for those participants who reported any use of alcohol at the 3 month follow-up (90 days from end of treatment; n=18) visit. Participants who did not report any alcohol use are not reported here.
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Groups:
- Mindfulness Based Relapse Prevention (MBRP): Women will receive the Mindfulness Based Relapse Prevention (MBRP) plus treatment as usual
  Mindfulness Based Relapse Prevention (MBRP): MBRP integrates coping skills from cognitive-behavioral relapse prevention therapy with Mindfulness Meditation (MM) practices, raising awareness of substance use triggers and reactive behavioral patterns, and teaching skillful coping responses.
- Treatment as Usual Only (TAU): Women will receive treatment as usual (less MBRP)
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Treatment as Usual Only (TAU)
Number analyzed (Participants) | 8 | 10
drinks per drinking day | 6.3 (5.7) | 6.6 (7.9)

9. Secondary Outcome: Time Line Follow Back (TLFB)
Description: Time Line Follow Back (TLFB) is a calendar based method that allows a clinician to obtain a quantitative amount of an individual's daily drinking during a given period of time. Participants are asked about the number of drinks they consumed on the days that they drank. The mean number of standard alcohol drinks per drinking day (DDD) for those participants who attended the 6 month follow-up visit who reported any drinking from the 3 month follow-up to the 6 month follow-up visit (n=20) is reported.
Time Frame: 6 month follow-up (90 days from the 3 month follow-up to the 6 month follow-up). Only those participants who reported any drinking at the 6 month follow-up visit are included (n=20).
Population: Participants who reported any drinking at the 6 month follow-up visit (90 days from 3 month to 6 month follow-up visit: n=20). Those who reported no drinking are not included here.
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Treatment as Usual Only (TAU)
Number analyzed (Participants) | 7 | 13
drinks per drinking day | 2.5 (1.7) | 3.7 (3.1)

10. Secondary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: The Five Factor Mindfulness Questionnaire (FFMQ) is a 24 item self report scale that measures the trait-like tendency to be mindful in daily life. It is comprised of aspects of mindfulness such as observing, describing, acting with awareness, non-judging, and non-reactivity. Item ratings range from 1 (never or very rarely true) to 5 (very often true or always true) and items are summed for a total score ranging from 0-120. Higher scores represent higher levels of mindfulness. Total scores for participants who attended the 8 week end of study visit (N=60) are reported here.
Time Frame: 8 week end of treatment visit (60 days baseline to end of treatment)
Population: Participants who attended the 8 week end of study visit (N=60) are reported/represented here. Not all participants attended end of treatment study visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
Number analyzed (Participants) | 32 | 28
score on a scale | 83.3 (3.1) | 78.4 (3.3)

11. Secondary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: The Five Factor Mindfulness Questionnaire (FFMQ) is a 24 item self report scale that measures the trait-like tendency to be mindful in daily life. It is comprised of aspects of mindfulness such as observing, describing, acting with awareness, non-judging, and non-reactivity. Item ratings range from 1 (never or very rarely true) to 5 (very often true or always true) and items are summed for a total score ranging from 0-120. Higher scores represent higher levels of mindfulness. Total scores for participants who attended the 3 month follow-up visit (n=53) are reported here.
Time Frame: 3 month follow-up (90 days from end of treatment to 3 month follow-up visit)
Population: Participants who attended the 3 month follow-up visit (N=53) are reported/represented here. Not all participants attended all study visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Treatment as Usual Only (TAU)
Number analyzed (Participants) | 26 | 27
score on a scale | 82.7 (3.4) | 79.4 (3.4)

12. Secondary Outcome: Five Factor Mindfulness Questionnaire (FFMQ)
Description: The Five Factor Mindfulness Questionnaire (FFMQ) is a 24 item self report scale that measures the trait-like tendency to be mindful in daily life. It is comprised of aspects of mindfulness such as observing, describing, acting with awareness, non-judging, and non-reactivity. Item ratings range from 1 (never or very rarely true) to 5 (very often true or always true) and items are summed for a total score ranging from 0-120. Higher scores represent higher levels of mindfulness. Total scores for participants who attended the 6 month follow-up visit (n=52) are reported here.
Time Frame: 6 month follow-up (90 days from 3 month follow-up visit to 6 month follow-up visit)
Population: Participants who attended the 6 month follow-up visit (N=52) are reported/represented here. Not all participants attended all study visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Treatment as Usual Only (TAU)
Number analyzed (Participants) | 25 | 27
score on a scale | 87.4 (3.5) | 79.3 (3.4)

13. Secondary Outcome: Difficulty in Emotion Regulation Scale (DERS)
Description: The Difficulty in Emotion Regulation Scale (DERS) is a 36-item self-report measure developed to assess clinically significant difficulties in emotion regulation. Responses range from 1 (almost never) to 5 (almost always) with higher scores indicating greater difficulties in emotion regulation. The range of scores is 0 to 180 and item scores are summed for a total score. Total scores for participants who attended the 8 week end of study visit (N=60) are reported here.
Time Frame: 8 week end of treatment (60 days baseline to end of treatment)
Population: Participants who attended the 8 week end of study visit (N=60) are reported/represented here. Not all participants attended all study visits.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Women Receiving MBRP Plus TAU: Women will receive the Mindfulness Based Relapse Prevention (MBRP) plus treatment as usual
  Mindfulness Based Relapse Prevention (MBRP): MBRP integrates coping skills from cognitive-behavioral relapse prevention therapy with Mindfulness Meditation (MM) practices, raising awareness of substance use triggers and reactive behavioral patterns, and teaching skillful coping responses.
- Women Receiving Treatment as Usual (TAU): Women will only receive treatment as usual (TAU less trauma focused group).
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving Treatment as Usual (TAU)
Number analyzed (Participants) | 32 | 28
score on a scale | 80.9 (4.8) | 85.7 (5.2)

14. Secondary Outcome: Difficulty in Emotional Regulation Scale (DERS)
Description: The Difficulty in Emotion Regulation Scale (DERS) is a 36-item self-report measure developed to assess clinically significant difficulties in emotion regulation. Responses range from 1 (almost never) to 5 (almost always) with higher scores indicating greater difficulties in emotion regulation. The range of scores is 0 to 180 and item scores are summed for a total score. Total scores for participants who attended the 3 month visit (N=53) are reported here.
Time Frame: 3 month follow-up (90 days end of treatment to 3 month follow-up)
Population: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Treatment as Usual Only (TAU)
Number analyzed (Participants) | 26 | 27
score on a scale | 85.4 (5.5) | 83.4 (5.4)

15. Secondary Outcome: Difficulty in Emotional Regulation Scale (DERS)
Description: The Difficulty in Emotion Regulation Scale (DERS) is a 36-item self-report measure developed to assess clinically significant difficulties in emotion regulation. Responses range from 1 (almost never) to 5 (almost always) with higher scores indicating greater difficulties in emotion regulation. The range of scores is 0 to 180 and item scores are summed for a total score. Total scores for participants who attended the 6 month visit (N=52) are reported here.
Time Frame: 6 month follow up (90 days from 3 month follow-up to 6 month follow-up)
Population: as for outcome 12
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention (MBRP) | Treatment as Usual Only (TAU)
Number analyzed (Participants) | 25 | 27
score on a scale | 76.4 (5.7) | 81.7 (5.4)

ADVERSE EVENTS:
Time Frame: Approximately 8-9 months
Arm/Group | Women Receiving MBRP Plus TAU | Women Receiving TAU
All-Cause Mortality (participants affected / at risk) | 0/45 | 1/45
Serious Adverse Events (participants affected / at risk) | 4/45 | 3/45
Other Adverse Events (participants affected / at risk) | 28/45 | 20/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Receiving MBRP Plus TAU (N=45) | Women Receiving TAU (N=45)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Knee Infection (Infections and infestations) | 1 (1) | 0 (0)
alcohol poisening (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Physical Assault (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — concussion, rib contusion, bruising, abrasions - overnight hospitalization
gall bladder stones (Hepatobiliary disorders) | 1 (1) | 0 (0) — Participant had a cholecystectomy
Severe opioid withdrawal (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Receiving MBRP Plus TAU (N=45) | Women Receiving TAU (N=45)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Cold (Infections and infestations) | 7 (7) | 5 (5)
Depressed mood (Psychiatric disorders) | 4 (4) | 3 (3)
Flu (Infections and infestations) | 5 (5) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 7 (7) | 5 (5)
Teeth Decay (Infections and infestations) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT02755103/Prot_SAP_000.pdf